CLINICAL TRIAL: NCT05116670
Title: Comparison of Care Practices, Mortality and Morbidity of Very Preterm Infants Between Two Tertiary Centers in Northwest and South of China
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhangbin Yu, Clinical Professor#Shenzhen People's Hospital, The Second Clinical Medical College of Jinan University
Other Study IDs: NMU-FY2021-58
Record Dates: First submitted 2021-10-31; First posted 2021-11-11 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Morality; Morbidity;Newborn; Very Preterm Maturity of Infant
Keywords: care practices; mortality; morbidity; very preterm infant; comparison

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qinghai Red Cross Hospital
- Shenzhen Baoan Women's and Children's Hospital

INTERVENTIONS:
Other:  — this is an observation study, no intervention is needed

SUMMARY:
Care practices, mortality and morbidity of very premature infants from two different tertiary centers were collected and compared, in order to discover areas for improvement where these two newborn centers can learn from each other.

DETAILED DESCRIPTION:
This retrospective cohort study was conducted in two hospitals,Qinghai Red Cross Hospital and Jinan University affiliated Shenzhen Baoan Women's and Children's Hospital.Very premature infants born with a gestational age between 22+0 - 31+6 weeks admitted to both centers during 3 years from January 1, 2018 to December 31, 2020 were studied. In both centers, data including maternal characteristics, neonatal characteristics, obstetric practices, delivery room practices, and neonatal outcomes, were collected by data abstractors in each NICU. Anonymous data was transferred to Shenzhen and analyses were performed at the newborn center of SZH.

ELIGIBILITY:
Inclusion Criteria:

* Very premature infants born with a gestational age between 22+0 - 31+6 weeks；
* Admitted to both centers during 3 years from January 1, 2018 to December 31, 2020.

Exclusion Criteria:

* Infants not born at QHH or SZH (out born);
* Infants who had major congenital anomalies;
* Infants admitted after 7 days of life.

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: Very premature infants born with a gestational age between 22+0 - 31+6 weeks admitted to newborn centers of Qinghai Red Cross Hospital and Shenzhen Baoan Women's and Children's Hospital from Jan 1, 2018 to Dec 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 807 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
mortality | Jan 1,2018 - Dec 31,2020
  death during hospitalisation and death after withdrawing treatment
Major morbidity | Jan 1,2018 - Dec 31,2020
  severe neurological injury, moderate to severe BPD, NEC or severe ROP

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Baoan Women's and Children's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided